CLINICAL TRIAL: NCT04158960
Title: Changes in Motor Skill Proficiency After Equine-Assisted Activities and Brain-Building Tasks in Youth With Neurodevelopmental Disorders
Brief Title: Motor Skill Proficiency After Equine-assisted Activities and Brain-building Tasks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Rhett Rigby, Associate Professor, Texas Woman's University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 17959
Record Dates: First submitted 2019-11-05; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Motor Delay; Motor Skills Disorders; Autism Spectrum Disorder; Attention Deficit Hyper Activity; Intellectual Disability; Sensory Disorders
MeSH Terms: conditions — Psychomotor Disorders; Motor Skills Disorders; Autism Spectrum Disorder; Intellectual Disability; Sensation Disorders

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Therapists were blinded to the outcome measures and assessments used to obtain those outcome measures in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Control period; no equine-assisted activities or brain-building activities occurred
- Equine-assisted activities period (Active Comparator): Period in which only equine-assisted activities were performed
  Interventions: Behavioral: Equine-assisted activities
- Washout (No Intervention): Washout period; no equine-assisted activities or brain-building activities occurred
- GaitWay period (Experimental): Period in which both equine-assisted activities and brain-building activities were performed
  Interventions: Behavioral: GaitWay program

INTERVENTIONS:
Behavioral: Equine-assisted activities — Participants performed riding-related activities on and off of a horse once per week for 8 weeks
  Other Names: EAA
  Arms: Equine-assisted activities period
Behavioral: GaitWay program — Participants performed riding-related activities on and off of a horse, along with brain-building activities including balance tasks, swinging, spinning, music therapy, and sensory tasks, all once per week for 8 weeks
  Other Names: GW
  Arms: GaitWay period

SUMMARY:
There is no current research to support the efficacy of a combination of equine-assisted activities (EAA) and brain building activities to influence motor skill competencies in youth with neurodevelopmental disorders (ND). The primary objective of this study was to quantify changes in motor skill proficiency before and after 8 weeks of EAA and brain-building activities in youth with ND. A secondary objective was to quantify changes in motor skill proficiency before and after 1 year of EAA and brain-building activities in youth with ND.

DETAILED DESCRIPTION:
Twenty-five youth completed the same 32-week protocol that was separated into 4, 8-week blocks, in the following order: a) control, b) EAA-only, c) washout, and d) GaitWay block (EAA and brain building activities). Before and after each block, motor skills were assessed using the Short Form of the Bruininks-Oseretsky Test of Motor Proficiency-Version 2 (BOT-2). Seven youth continued with the GaitWay intervention for one additional year, and the BOT-2 Short Form was also administered following this intervention. A repeated-measures analysis-of-variance was performed to compare BOT-2 subtest and overall scores between interventions. A significance of .05 was used. Manual dexterity was higher at Post-Washout versus Pre-Control (p = .018) and Post-Control (p = .024), and at Post-GaitWay versus Pre-Control (p = .037). Upper-limb coordination was higher Post-GaitWay versus Post-Control (p = .050). When compared to Pre-Control, strength was higher at Post-EAA (p = .028) and at Post-GaitWay (p = .015). Overall scores were higher at Post-GaitWay when compared to Pre-Control (p = .003) and Post-Control (p = .009). Among the seven participants who participated in the 1-year follow-up GaitWay motor skills were maintained for one year following the Post-GaitWay testing session. A combination of EAA and brain building activities may be an effective therapeutic modality to improve and maintain motor skill proficiency in youth with ND.

ELIGIBILITY:
Inclusion Criteria:

* age 5 to 18 years
* diagnosis of a neurodevelopmental disorder (as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5))
* had the ability to follow verbal directions,
* Clearance to participate from a medical professional

Exclusion Criteria:

* a perfect score on the motor proficiency test at the first testing session
* presence of seizures within the past 6 months controlled by medication
* a known allergy to horses
* any surgical procedures performed within the 6 months
* regular horseback riding experience of any kind during the past year

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Fine motor precision | 0-5 minutes
  Subtest #1 on the Bruininks-Oseretsky Test of Motor Proficiency (Version 2) Short Form. Tasks include drawing through lines, folding paper. Each task within this subtest is scored on a scale from 0-7 (with 7 representing the best outcome).
Fine motor integration | 0-5 minutes
  Subtest #2 on the Bruininks-Oseretsky Test of Motor Proficiency (Version 2) Short Form. Task includes copying a star and a square. The task within this subtest is scored on a scale from 0-5 (with 5 representing the best outcome).
Manual dexterity | 15 seconds
  Subtest #3 on the Bruininks-Oseretsky Test of Motor Proficiency (Version 2) Short Form. Task includes transferring pennies. The task within this subtest is scored on a scale from 0-9 (with 9 representing the best outcome).
Bilateral coordination | 0-5 minutes
  Subtest #4 on the Bruininks-Oseretsky Test of Motor Proficiency (Version 2) Short Form. Tasks include jumping in place with arms and legs on same side of the body synchronized, and tapping feet and fingers simultaneously, with hands and feet on the same side of the body synchronized. The jumping task within this subtest is scored on a scale from 0-3 (with 3 representing the best outcome). The tapping task within this subtest is scored on a scale from 0-4 (with 4 representing the best outcome).
Balance | 1 minute
  Subtest #5 on the Bruininks-Oseretsky Test of Motor Proficiency (Version 2) Short Form. Tasks include walking forward on a line, standing on one leg on a balance beam with eyes open. Each task within this subtest is scored on a scale from 0-4 (with 4 representing the best outcome).
Running speed and agility | 15 seconds
  Subtest #6 on the Bruininks-Oseretsky Test of Motor Proficiency (Version 2) Short Form. Task includes one-legged stationary hop. The task within this subtest is scored on a scale from 0-10 (with 10 representing the best outcome).
Upper-limb coordination | 0-5 minutes
  Subtest #7 on the Bruininks-Oseretsky Test of Motor Proficiency (Version 2) Short Form. Tasks include dropping and catching a ball with both hands, dribbling a ball with alternating hands. The dropping and catching task within this subtest is scored on a scale from 0-5 (with 5 representing the best outcome). The dribbling task within this subtest is scored on a scale from 0-7 (with 7 representing the best outcome).
Strength | 1 minute
  Subtest #8 on the Bruininks-Oseretsky Test of Motor Proficiency (Version 2) Short Form. Tasks include knee push-ups and sit-ups. Each task within this subtest is scored on a scale from 0-10 (with 10 representing the best outcome).
Overall Motor Skill Scores | 2 minutes
  Sum of all scores from the 8 subtests of the Bruininks-Oseretsky Test of Motor Proficiency (Version 2) Short Form. Total scores can range from 0-88 (with 88 representing the best outcome)

SECONDARY OUTCOMES:
Caregiver reports | 5 minutes
  Anecdotal reports from caregivers regarding progress of the participant

CONTACTS AND LOCATIONS:
Overall Officials: Brandon R Rigby, PhD, Principal Investigator — Texas Woman's University

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) may be shared by contacting the corresponding author for the study once it is published. All data related to motor skill tasks, including fine motor precision, fine motor integration, manual dexterity, bilateral coordination, balance, running speed and agility, upper-limb coordination, strength, and overall motor skill scores may be shared upon request.

REFERENCES:
- [Derived] Rigby BR, Davis RW, Bittner MD, Harwell RW, Leek EJ, Johnson GA, Nichols DL. Changes in Motor Skill Proficiency After Equine-Assisted Activities and Brain-Building Tasks in Youth With Neurodevelopmental Disorders. Front Vet Sci. 2020 Jan 31;7:22. doi: 10.3389/fvets.2020.00022. eCollection 2020. PMID 32083104